CLINICAL TRIAL: NCT04739280
Title: Women's Assessed Cardiovascular Evaluation With MCG
Acronym: WACE-MCG
Status: Completed | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1000-1
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Ischemia; Cardiac Disease; Risk Factor, Cardiovascular
Keywords: Cardiovascular Disease; Magnetic Field Map; CardioFLux; Ischemia; Magnetocardiography; MCG
MeSH Terms: conditions — Ischemia; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single center registry for WACE: We propose a single center registry for patients requiring diagnostic, screening, or surveillance for potential or existing cardiac illness. All eligible patients will undergo an MCG with periodic follow-ups. No treatment decisions will be based on the MCG findings, until CardioFlux has appropriate FDA labelling for clinical use.
  Interventions: Device: CardioFlux Magnetocardiography

INTERVENTIONS:
Device: CardioFlux Magnetocardiography — Magnetocardiography

SUMMARY:
Cardiovascular disease (CVD) is the number one cause of death for women over the age of 25, accounting for 1 of every 3 female deaths. Research has shown that while hypertension in women is less controlled, they are also less likely to be identified with ischemic heart disease and when diagnosed treated less aggressively than men. Moreover, women who are diagnosed with breast cancer have an increased risk for cardiovascular disease. The Women's Assessed Cardiovascular Evaluation with MCG (WACE-MCG) study is designed to collect CardioFlux scans on a select group of female volunteers who are Ms. Medicine patients. CardioFlux is used as a noninvasive MCG tool that analyzes and records the magnetic fields of the heart to detect various forms of heart disease. There will be a 12-month duration of the study where we propose to collect screening data from approximately 200 volunteers who present to the Genetesis facility for a 5-minute CardioFlux MCG scan. The volunteers will be contacted at intervals over a 1-year period for follow-up data and may choose whether or not they would like to provide follow-up data or participate in another scan.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years of age at the time of enrollment. Female Patients deemed at risk for cardiovascular disease (breast cancer survivors, patients referred to cardiologists, prior COVID-19 patients, etc.)

Exclusion Criteria:

< 18 years of age Patients unable to fit into device Non-ambulatory patients Positive response on CardioFlux Pre-Screening Form Patients with claustrophobia or unable to lie supine for 5 minutes Pregnant women Poor candidate for follow-up (e.g. no access to phone) Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must identify as Female
Study Population: The following describes the targeted population population
  ≥ 18 years of age at the time of enrollment. Female Patients deemed at risk for cardiovascular disease (breast cancer survivors, patients referred to cardiologists, prior COVID-19 patients, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Accuracy Statistics | 6 Months
  analyzing the accuracy of CardioFlux
Specificity Statistics | 6 months
  analyzing the specificity of CardioFlux

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Senagore, M.D., Principal Investigator — Genetesis Inc.
Locations (1):
- Genetesis Facility, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duda-Pyszny D, Trzeciak P, Gasior M. Coronary artery disease in women. Kardiochir Torakochirurgia Pol. 2018 Mar;15(1):44-48. doi: 10.5114/kitp.2018.74675. Epub 2018 Mar 28. PMID 29681961
- [Background] Garcia M, Mulvagh SL, Merz CN, Buring JE, Manson JE. Cardiovascular Disease in Women: Clinical Perspectives. Circ Res. 2016 Apr 15;118(8):1273-93. doi: 10.1161/CIRCRESAHA.116.307547. PMID 27081110
- [Background] Merz CN, Kelsey SF, Pepine CJ, Reichek N, Reis SE, Rogers WJ, Sharaf BL, Sopko G. The Women's Ischemia Syndrome Evaluation (WISE) study: protocol design, methodology and feasibility report. J Am Coll Cardiol. 1999 May;33(6):1453-61. doi: 10.1016/s0735-1097(99)00082-0. PMID 10334408
- [Background] Baldassarre LA, Raman SV, Min JK, Mieres JH, Gulati M, Wenger NK, Marwick TH, Bucciarelli-Ducci C, Bairey Merz CN, Itchhaporia D, Ferdinand KC, Pepine CJ, Walsh MN, Narula J, Shaw LJ; American College of Cardiology's Cardiovascular Disease in Women Committee. Noninvasive Imaging to Evaluate Women With Stable Ischemic Heart Disease. JACC Cardiovasc Imaging. 2016 Apr;9(4):421-35. doi: 10.1016/j.jcmg.2016.01.004. PMID 27056162
- [Background] Barish R, Lynce F, Unger K, Barac A. Management of Cardiovascular Disease in Women With Breast Cancer. Circulation. 2019 Feb 19;139(8):1110-1120. doi: 10.1161/CIRCULATIONAHA.118.039371. PMID 30779651
- [Background] Chaikovsky I, Hailer B, Sosnytskyy V, Lutay M, Mjasnikov G, Kazmirchuk A, Bydnyk M, Lomakovskyy A, Sosnytskaja T. Predictive value of the complex magnetocardiographic index in patients with intermediate pretest probability of chronic coronary artery disease: results of a two-center study. Coron Artery Dis. 2014 Sep;25(6):474-84. doi: 10.1097/MCA.0000000000000107. PMID 24667125
- [Background] Goernig M, Liehr M, Tute C, Schlosser M, Haueisen J, Figulla HR, Leder U. Magnetocardiography based spatiotemporal correlation analysis is superior to conventional ECG analysis for identifying myocardial injury. Ann Biomed Eng. 2009 Jan;37(1):107-11. doi: 10.1007/s10439-008-9598-5. Epub 2008 Nov 18. PMID 19015988
- [Background] Hailer B, Chaikovsky I, Auth-Eisernitz S, Schafer H, Van Leeuwen P. The value of magnetocardiography in patients with and without relevant stenoses of the coronary arteries using an unshielded system. Pacing Clin Electrophysiol. 2005 Jan;28(1):8-16. doi: 10.1111/j.1540-8159.2005.09318.x. PMID 15660796
- See also: Women & Cardiovascular Disease — http://my.clevelandclinic.org/health/diseases/17645-women--cardiovascular-disease